CLINICAL TRIAL: NCT01606189
Title: A Double Blind, Randomised, Three Way Crossover Study Comparing Two Different Sublingual Cannabis Based Medicine Extracts With Placebo, in Patients With Chronic Pain Due to Brachial Plexus Injury.
Brief Title: A Study to Compare Sublingual Cannabis Based Medicine Extracts With Placebo to Treat Brachial Plexus Injury Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWBP0101
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GW-1000-02 (Experimental): Active treatment.
  Interventions: Drug: GW-1000-02
- GW-2000-02 (Experimental): Active treatment.
  Interventions: Drug: GW-2000-02
- Placebo (Placebo Comparator): Placebo control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW-1000-02 — Contains delta-9-tetrahydrocannabinol (THC) (25 mg/ml) and cannabidiol (CBD) (25mg/ml) as extract of Cannabis sativa L, with peppermint oil, 0.05% (v/v), in ethanol:propylene glycol (50:50) excipient. Each actuation delivered 100 μl (THC 2.5 mg and CBD 2.5 mg). The maximum daily exposure was set at 48 actuations per day.
  Other Names: Sativex
  Arms: GW-1000-02
Drug: GW-2000-02 — Contains THC (25 mg/ml) as extract of Cannabis sativa L, with peppermint oil, 0.05% (v/v), in ethanol:propylene glycol (50:50) excipient. Each actuation delivered 100 μl (THC 2.5 mg). The maximum daily exposure was set at 48 actuations per day.
  Arms: GW-2000-02
Drug: Placebo — Contains peppermint oil, 0.05% (v/v), quinoline yellow, 0.005% (w/v), sunset yellow, 0.0025% (w/v), in ethanol:propylene glycol (50:50) excipient. Each actuation delivered 100 μl. The maximum daily exposure was set at 48 actuations per day.
  Arms: Placebo

SUMMARY:
A study to compare the efficacy of two sublingual cannabinoid based medicine extracts with placebo in the treatment of chronic pain due to brachial plexus injury.

DETAILED DESCRIPTION:
This study used a three way crossover study design. Eligible patients recorded their symptoms during a one to two week baseline period, then entered a three period, double blind, randomised crossover of GW-1000-02, GW-2000-02 and placebo. Each period lasted two weeks, with no washout between periods. There were six possible treatment sequences. The primary analysis was based on Box Scale-11 pain severity scores recorded throughout the study in patient daily diary booklets. Blood samples were taken from patient-volunteers at the beginning of each period, for measurement of plasma cannabinoid concentration.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above.
* Brachial plexus pain, at least 18 months after the initial injury.
* Reported weekly brachial plexus pain at the required severity at Visits 1 and 2; a Box Scale-11 pain severity score of four boxes or above.
* A pattern of pain that in the Investigator's opinion had been stable during the four weeks before study entry.
* Stable regular medication during the four weeks before study entry.
* A maximum tricyclic antidepressant dose of 75 mg per day, if applicable.
* No cannabinoid use (cannabis, Marinol® or Nabilone) at least seven days before study entry or during the study.
* If sexually active; was either using effective contraception during the study and for three months thereafter or had been surgically sterilised or, if female, was post-menopausal. All patients agreed to use a barrier method of contraception in addition to their usual form of oral or depot contraception.
* Willing and able to undertake and comply with all study requirements.
* Willing and able to consider and understand the patient information leaflet and consent form and to give informed consent. Those patients unable to read or to sign the document were managed as detailed in the Declaration of Helsinki.
* Willing for his or her general practitioner, and consultant if appropriate, to be informed of study participation.
* Willing for his or her name to be notified to Home Office for participation in the study.

Exclusion Criteria:

* Abuse or strong suspicion of drug abuse, including alcohol or cannabis, or in the investigator's opinion had a tendency to drug dependency or substance abuse. Patients with a history of abuse could have been included at the discretion of the investigator.
* Known or suspected adverse reaction to cannabinoids.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medication.
* History of any type of schizophrenia, any other psychotic illness, or other significant psychiatric illness other than depression associated with chronic illness.
* Regular levodopa therapy (Sinemet®, Sinemet plus®, Levodopa®, L-dopa®, Madopar®, Benserazide®) within seven days of study entry.
* Serious cardiovascular disorder including recent angina, uncontrolled hypertension or an uncontrolled symptomatic cardiac arrhythmia.
* History of significant renal or hepatic impairment as shown in medical history or indicated by clinical laboratory results from samples.
* History of active epilepsy or convulsions.
* Nerve surgery within six months of study entry or any other surgery within two months of study entry.
* Elective surgery, other procedures requiring general anaesthesia, or a planned hospital admission that would have taken place during the study, other than a hospital admission under the care of the study investigator.
* Terminal illness.
* Pregnancy, lactation or expected non-compliance with the contraceptive measures called for by the protocol.
* Participation in any other pharmacological clinical research study in the 12 weeks before study entry.
* Planned travel outside the UK between study entry and the end of the crossover phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-12; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal National Orthopaedic Hospital, Middlesex, United Kingdom

REFERENCES:
- [Result] Berman JS, Symonds C, Birch R. Efficacy of two cannabis based medicinal extracts for relief of central neuropathic pain from brachial plexus avulsion: results of a randomised controlled trial. Pain. 2004 Dec;112(3):299-306. doi: 10.1016/j.pain.2004.09.013. PMID 15561385

RESULTS

PARTICIPANT FLOW:
Groups:
- GW-1000-02 First, Then GW-2000-02, Then Placebo: GW-1000-02 first (14-20 days), then GW-2000-02 (14-20 days), then placebo (14-20 days).
  Each actuation of GW-1000-02 delivered a dose containing 2.5 mg THC and 2.5 mg CBD, each actuation of GW-2000-02 delivered a dose containing 2.5 mg THC and each actuation of placebo delivered the excipients only. Patients were required to take no more than eight actuations of study medication within each three hour period, and no more than 48 actuations each day (24 hour period).
- GW-2000-02 First, Then GW-1000-02, Then Placebo; GW-2000-02 First, Then Placebo, Then GW-1000-02: GW-2000-02 first (14-20 days), then GW-1000-02 (14-20 days), then placebo (14-20 days).
  Each actuation of GW-1000-02 delivered a dose containing 2.5 mg THC and 2.5 mg CBD, each actuation of GW-2000-02 delivered a dose containing 2.5 mg THC and each actuation of placebo delivered the excipients only. Patients were required to take no more than eight actuations of study medication within each three hour period, and no more than 48 actuations each day (24 hour period).
- Placebo First, Then GW-1000-02, Then GW-2000-02; Placebo First, Then GW-2000-02, Then GW-1000-02: Placebo first (14-20 days), then GW-1000-02 (14-20 days), then GW-2000-02 (14-20 days).
  Each actuation of GW-1000-02 delivered a dose containing 2.5 mg THC and 2.5 mg CBD, each actuation of GW-2000-02 delivered a dose containing 2.5 mg THC and each actuation of placebo delivered the excipients only. Patients were required to take no more than eight actuations of study medication within each three hour period, and no more than 48 actuations each day (24 hour period).
- GW-1000-02 First, Then Placebo, Then GW-2000-02: GW-1000-02 first (14-20 days), then placebo (14-20 days), then GW-2000-02 (14-20 days).
  Each actuation of GW-1000-02 delivered a dose containing 2.5 mg THC and 2.5 mg CBD, each actuation of GW-2000-02 delivered a dose containing 2.5 mg THC and each actuation of placebo delivered the excipients only. Patients were required to take no more than eight actuations of study medication within each three hour period, and no more than 48 actuations each day (24 hour period).
Period: First Intenvention (14-20 Days)
Arm/Group | GW-1000-02 First, Then GW-2000-02, Then Placebo | GW-2000-02 First, Then GW-1000-02, Then Placebo | Placebo First, Then GW-1000-02, Then GW-2000-02 | GW-1000-02 First, Then Placebo, Then GW-2000-02 | Placebo First, Then GW-2000-02, Then GW-1000-02 | GW-2000-02 First, Then Placebo, Then GW-1000-02
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intenvention (14-20 Days)
Arm/Group | GW-1000-02 First, Then GW-2000-02, Then Placebo | GW-2000-02 First, Then GW-1000-02, Then Placebo | Placebo First, Then GW-1000-02, Then GW-2000-02 | GW-1000-02 First, Then Placebo, Then GW-2000-02 | Placebo First, Then GW-2000-02, Then GW-1000-02 | GW-2000-02 First, Then Placebo, Then GW-1000-02
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Third Intenvention (14-20 Days)
Arm/Group | GW-1000-02 First, Then GW-2000-02, Then Placebo | GW-2000-02 First, Then GW-1000-02, Then Placebo | Placebo First, Then GW-1000-02, Then GW-2000-02 | GW-1000-02 First, Then Placebo, Then GW-2000-02 | Placebo First, Then GW-2000-02, Then GW-1000-02 | GW-2000-02 First, Then Placebo, Then GW-1000-02
Started | 8 | 8 | 8 | 8 | 8 | 7
Completed | 8 | 8 | 8 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: GW-1000-02, GW-2000-02 and Placebo: As this was a crossover study design, all patients were to receive all study treatments: GW-1000-02, GW-2000-02 and placebo.
Arm/Group | All Study Treatments: GW-1000-02, GW-2000-02 and Placebo
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.53 (10.342)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 46
Region of Enrollment [Number; unit: participants]
  United Kingdom | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Box Scale-11 Pain Review Score at the End of Each Treatment Period (Each Lasting 14-20 Days)
Description: Each day patients recorded in their patient diary, the severity of their pain during the previous 24 hours using a Box Scale-11 pain score ranging from zero "no pain at all" to 10 "pain as bad as you can imagine". The Box Scale-11 pain score endpoint for each assessment period was the average of all available data recorded during the seven whole days prior to the visit immediately subsequent to that period, but only including data from Day 8 onwards. A negative value indicates an improvement in pain score from baseline.
Time Frame: Up to 74 days
Population: All patients who entered the study, were randomised and had some on-treatment efficacy data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GW-1000-02: Each 100 micro litre actuation contains THC (25 mg/ml) and CBD (25mg/ml). The maximum dose allowed was 48 actuations (130 mg THC and 120 mg CBD) per 24 hours.
- GW-2000-02: Each 100 micro litre actuation contains THC (25 mg/ml). The maximum dose allowed was 48 actuations (130 mg THC) per 24 hours.
- Placebo: Contains no active drug but colourants and excipients. Maximum permitted dose was 48 actuations in 24 hours.
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 45 | 47 | 47
units on a scale | -0.6 (1.13) | -0.6 (1.34) | 0.0 (1.23)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Box Scale-11 pain scores were compared between treatment groups using an analysis of variance (ANOVA). The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Box Scale-11 Pain Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.005, ANOVA; Estimated mean treatment difference = -0.58, 95% CI 2-sided [-0.98 to -0.18]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; Box Scale-11 pain scores were compared between treatment groups using an ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Box Scale-11 Pain Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.002, ANOVA; Estimated mean treatment difference = -0.64, 95% CI 2-sided [-1.03 to -0.24]

2. Secondary Outcome: Change From Baseline in the Mean Sleep Disturbance Score at the End of Each Treatment Period (Each Lasting 14-20 Days).
Description: Each day patients recorded in their patient diary the number of times they were woken due to pain during the previous night. The results were recorded as "None", "Once", "Twice" and "More Than Twice" and converted to a four point scale, zero to three respectively. The treatment days and the assessment periods were defined in the same way as for the Box Scale-11 pain score. A negative value indicates an improvement from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 44 | 46 | 46
units on a scale | -0.2 (0.43) | -0.4 (0.51) | 0.0 (0.47)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Sleep disturbance scores were compared between treatment groups using ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Sleep disturbance Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.017, ANOVA; Estimated mean treatment difference = -0.20, 95% CI 2-sided [-0.37 to -0.04]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Estimated mean treatment difference = -0.33, 95% CI 2-sided [-0.49 to -0.16]

3. Secondary Outcome: Change From Baseline in the Mean Box Scale-11 Sleep Quality Score at the End of Each Treatment Period (Each Lasting 14-20 Days).
Description: Each day patients recorded in their patient diary the quality of their sleep during the previous night using a Box Scale-11 sleep score ranging from zero "Worst Imaginable" to 10 "Best Imaginable". The treatment days and the assessment periods were defined in the same way as for the Box Scale-11 pain score. A positive value indicates an improvement from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 45 | 47 | 47
units on a scale | 0.9 (1.22) | 1.2 (1.39) | 0.4 (1.40)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Sleep quality scores were compared between treatment groups using ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Sleep Quality Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.019, ANOVA; Estimated mean treatment difference = 0.55, 95% CI 2-sided [0.09 to 1.01]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.001, ANOVA; Estimated mean treatment difference = 0.79, 95% CI 2-sided [0.33 to 1.24]

4. Secondary Outcome: Change From Baseline in the Mean McGill Pain Questionnaire Part 1 Score for 'Total Pain Intensity' at the End of Each Treatment Period (Each Lasting 14-20 Days)
Description: Part 1 of the questionnaire related to the intensity of 15 different types of pain. Intensity was recorded separately for each type of pain on a zero to three scale, where zero = "None", one = "Mild", two = "Moderate" and three = "Severe". The total intensity was defined as the unweighted sum of the 15 scores, giving a minimum possible score of zero (lowest pain score) and a maximum possible score of 45 (highest pain score). The distribution of each of the 15 types of pain was summarised at baseline and for each treatment. A negative value indicates an improvement in pain from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 46 | 46 | 48
units on a scale | -3.2 (8.91) | -3.8 (9.37) | -1.8 (9.26)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Total pain intensity scores were compared between treatment groups using ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Total Pain Intensity Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.146, ANOVA; Estimated mean treatment difference = -1.55, 95% CI 2-sided [-3.64 to 0.55]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.040, ANOVA; Estimated mean treatment difference = -2.20, 95% CI 2-sided [-4.29 to -0.10]

5. Secondary Outcome: Change From Baseline in the Mean McGill Pain Questionnaire Part 2 Score for 'Intensity of Pain' at the End of Each Treatment Period (Each Lasting 14-20 Days)
Description: Part 2 of the questionnaire recorded the intensity of pain at present. Results were recorded on a VAS ranging from zero "No pain" to 100 "Worst possible pain". Intensity of pain was summarised and analysed in the same manner as the primary efficacy parameter of Box Scale-11 pain score. A negative value indicates an improvement from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 46 | 47 | 48
units on a scale | -14.9 (25.15) | -17.3 (26.74) | -8.0 (26.92)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Intensity of Pain scores were compared between treatment groups using ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Intensity of Pain Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.092, ANOVA; Estimated mean treatment difference = -7.28, 95% CI 2-sided [-15.78 to 1.21]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.037, ANOVA; Estimated mean treatment difference = -8.99, 95% CI 2-sided [-17.41 to -0.57]

6. Secondary Outcome: Change From Baseline in the Number of Patients Who Reported 'No Pain' or 'Mild Pain' Using a McGill Pain Questionnaire Part 3 Score for 'Strength of Pain at Present' at the End of Each Treatment Period (Each Lasting 14-20 Days)
Description: Part 3 of the questionnaire recorded the strength of pain at present. Results were recorded in six categories which were classified as "No Pain", "Mild", "Discomforting", "Distressing", "Horrible" and "Excruciating". The change from baseline in the number of patients who reported "No Pain" or "Mild Pain" at the end of the respective treatment periods is presented. An increase in number indicates an improvement from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 46 | 47 | 48
participants | 4 | 4 | 3
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Pain at present was analysed using the Mann-Whitney test with a correction for ties. Results were presented in terms of the sums of the ranks for the two groups, the Mann-Whitney U statistic and the associated p-value; Test type: Superiority or Other; p = 0.328, Wilcoxon (Mann-Whitney); Mann-Whitney U statistic = 1222.0
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.560, Wilcoxon (Mann-Whitney); Mann-Whitney U statistic = 1200.5

7. Secondary Outcome: Change From Baseline in the Mean Pain Disability Index Score at the End of Each Treatment Period (Each Lasting 14-20 Days).
Description: The Pain Disability Index consisted of seven assessments representing different aspects of disability due to pain. Each assessment was scored on a zero to 10 scale, where zero equated with "no disability" and 10 equated with "total disability". The total Pain Disability Index score was the unweighted sum of the seven pain scores, ranging from zero to 70. A negative value indicates an improvement from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 46 | 47 | 48
units on a scale | -5.3 (9.97) | -3.1 (10.37) | -3.6 (7.69)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; Pain Disability Index scores were compared between treatment groups using ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: Pain Disability Index Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.181, ANOVA; Estimated mean treatment difference = -1.75, 95% CI 2-sided [-4.32 to 0.83]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.739, ANOVA; Estimated mean treatment difference = 0.43, 95% CI 2-sided [-2.12 to 2.98]

8. Secondary Outcome: Change From Baseline in the Mean 12-Item General Health Questionnaire Score at the End of Each Treatment Period (Each Lasting 14-20 Days).
Description: The 12-Item General Health Questionnaire consisted of 12 general health questions. Each question was scored on a zero to three scale, where zero represented the better assessment. The total score was the unweighted sum of the 12 scores, ranging from zero to 36. A negative value indicates an improvement from baseline.
Time Frame: Up to 74 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 46 | 47 | 48
units on a scale | -2.2 (6.70) | -1.2 (6.12) | 0.1 (3.92)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; 12-Item General Health Questionnaire scores were compared between treatment groups using ANOVA. The model included factors for patient, treatment and period. The significance of the overall treatment effect was assessed using the F-test from the ANOVA. The model used was as follows: 12-Item General Health Questionnaire Score = Patient + Treatment + Period; Test type: Superiority or Other; p = 0.015, ANOVA; Estimated mean treatment difference = -2.23, 95% CI 2-sided [-4.01 to -0.45]
Statistical Analysis 2: Comparison: GW-2000-02 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.178, ANOVA; Estimated mean treatment difference = -1.21, 95% CI 2-sided [-2.97 to 0.56]

9. Secondary Outcome: Incidence of Adverse Events as a Measure of Patient Safety.
Description: The number of patients who experienced an adverse event during the course of study is presented.
Time Frame: Up to 114 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Number analyzed (Participants) | 46 | 47 | 48
participants | 34 | 37 | 20

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the study onset to up to 40 days follow-up (up to 114 days) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | GW-1000-02 | GW-2000-02 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 34/46 | 37/47 | 20/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=46) | GW-2000-02 (N=47) | Placebo (N=48)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=46) | GW-2000-02 (N=47) | Placebo (N=48)
Dizziness (Nervous system disorders) | 9 | 11 | 4
Somnolence (Nervous system disorders) | 7 | 6 | 5
Dysgeusia (Nervous system disorders) | 10 | 5 | 0
Headache Not Otherwise Specified (Nervous system disorders) | 0 | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 3
Dry Mouth (Nervous system disorders) | 3 | 3 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 4
Feeling Drunk (General disorders) | 4 | 4 | 0
Lethargy (General disorders) | 0 | 3 | 0
Pain Exacerbated (General disorders) | 0 | 4 | 0
Thirst (General disorders) | 0 | 3 | 0
Euphoric Mood (Psychiatric disorders) | 3 | 2 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 0
Paresthesia Oral (Nervous system disorders) | 0 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 2 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 2 | 0
Panic Attack (Psychiatric disorders) | 0 | 2 | 0
Appetite Increased (Metabolism and nutrition disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.